CLINICAL TRIAL: NCT04778410
Title: A Phase 2 Multi-Arm Study of Magrolimab Combinations in Patients With Myeloid Malignancies
Brief Title: Study of Magrolimab Combinations in Participants With Myeloid Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate the study.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-546-5920; 2021-003833-13 (EudraCT Number)
Expanded Access: NCT05627466 (No longer available)
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Myeloid Malignancies
MeSH Terms: interventions — magrolimab; Azacitidine; venetoclax; Mitoxantrone; Etoposide; Cytarabine; cc-486

STUDY DESIGN:
Intervention Model Description: After completion of Safety Run-in cohorts and identification of the RP2D for the specific cohorts, participants may be enrolled to the corresponding Phase 2 cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (1L Unfit AML): Magrolimab + Venetoclax + Azacitidine (Experimental): Participants with newly diagnosed untreated acute myeloid leukemia (AML) who are ineligible for intensive induction chemotherapy will receive magrolimab 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then every week (QW) x 5 doses; 30 mg/kg every 2 weeks (Q2W) beginning 1 week after the 5 weekly 30 mg/kg dose in every 28-day cycle along with azacitidine and venetoclax first in the Safety Run-in Cohort. Once the safety of recommended dose of magrolimab is confirmed, the participants in Phase 2 Cohort will be enrolled to receive the treatment.
  Interventions: Drug: Magrolimab; Drug: Azacitidine; Drug: Venetoclax
- Cohort 2 (R/R AML): Magrolimab + Mitoxantrone + Etoposide + Cytarabine (Experimental): Participants with relapsed/refractory (RR) AML after intensive induction chemotherapy will receive magrolimab 1 mg/ on Days 1, 4; 15 mg/kg, on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 doses; 30 mg/kg Q2W beginning 1 week after the 5 weekly 30 mg/kg dose along with mitoxantrone + etoposide + cytarabine (MEC) first in the Safety Run-in Cohort. Once the safety of recommended dose of magrolimab is confirmed, the participants in Phase 2 Cohort will be enrolled to receive the treatment.
  Interventions: Drug: Magrolimab; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine
- Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486 (Experimental): Participants with AML who achieved CR or CRi with MRD positivity following intensive induction chemotherapy will receive magrolimab 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 doses; 30 mg/kg Q2W beginning 1 week after the 5 weekly 30 mg/kg dose along with CC-486 as maintenance therapy first in the Safety Run-in Cohort. Once the safety of recommended dose of magrolimab is confirmed, the participants in Phase 2 Cohort will be enrolled to receive the treatment.
  Interventions: Drug: Magrolimab; Drug: CC-486

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously
  Other Names: GS-4721
Drug: Azacitidine — Administered either subcutaneously or IV, 75 mg/milligram per square (m^2) on Days 1 to 7 or Days 1 to 5, 8 and 9 during every cycle
  Arms: Cohort 1 (1L Unfit AML): Magrolimab + Venetoclax + Azacitidine
Drug: Venetoclax — Administered orally at a dose of 100 mg on Day 1, 200 mg on Day 2, 400 mg on Days 3-28 during Cycle 1, followed by 400 mg on Days 1-28 during every cycle
  Arms: Cohort 1 (1L Unfit AML): Magrolimab + Venetoclax + Azacitidine
Drug: Mitoxantrone — Administered intravenously, 8 mg/m^2 on Days 1-5 during Cycle 1 to Cycle 3
  Arms: Cohort 2 (R/R AML): Magrolimab + Mitoxantrone + Etoposide + Cytarabine
Drug: Etoposide — Administered intravenously, 100 mg/m^2 on Days 1-5 during Cycle 1 to Cycle 3
  Arms: Cohort 2 (R/R AML): Magrolimab + Mitoxantrone + Etoposide + Cytarabine
Drug: Cytarabine — Administered intravenously, 1000 mg/m^2 on Days 1-5 during Cycle 1 to Cycle 3
  Arms: Cohort 2 (R/R AML): Magrolimab + Mitoxantrone + Etoposide + Cytarabine
Drug: CC-486 — Administered orally, 300 mg on Days 1-14 during each cycle
  Other Names: Onureg
  Arms: Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486

SUMMARY:
The goal of this clinical study is to learn more about the safety and dosing of the study drug, magrolimab (Mag), in combination with anti-leukemia therapies in participants with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
The anti-leukemia therapies are defined as follows:

* Venetoclax (Ven)
* Azacitidine (Aza)
* Mitoxantrone, etoposide, and cytarabine (MEC)

This study consists of 3 safety run-in cohorts;

* Safety Run-in Cohort 1 (1L Unfit AML Mag + Ven + Aza)
* Safety Run-in Cohort 2 (R/R AML Mag + MEC)
* Safety Run-in Cohort 3 (Post-chemo Maintenance Mag + CC-486)

Participants will receive treatment at the assigned dose level for at least 4 cycles in the Safety Run-in cohorts, after which they may continue at the assigned dose level or switch to the RP2D upon agreement between the investigator and the sponsor. After completion of each safety run-in cohort and identification of the RP2D for that cohort, participants may be enrolled into the corresponding Phase 2 cohorts;

* Phase 2 Cohort 1 (1L Unfit AML Mag + Ven + Aza)
* Phase 2 Cohort 2 (R/R AML Mag + MEC)
* Phase 2 Cohort 3 (Post-chemo Maintenance Mag + CC-486)

Cycle length is 28 days for both the Safety Run-in and Phase 2 cohorts.

Note: All cohorts are closed to screening and enrollment.

ELIGIBILITY:
Key Inclusion Criteria:

All Individuals:

* White blood cell (WBC) count ≤ 20 × 10^3/microliter (μL) prior to first dose of study treatment. If the individual's WBC count is > 20 × 10^3/ μL prior to first dose of study treatment, the individual can be enrolled, assuming all other eligibility criteria are met
* For individuals with prior cardiac history, the hemoglobin must be ≥ 9 grams per deciliter (g/dL) prior to initial dose of study treatment. Transfusions are allowed to meet hemoglobin eligibility
* Adequate liver function
* Adequate renal function
* Individual has provided informed consent
* Individual is willing and able to comply with clinic visits and procedures outlined in the study protocol
* Pretreatment blood cross-match completed
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol- specified method(s) of contraception
* Individuals must be willing to consent to mandatory pretreatment and on-treatment bone marrow biopsies (trephines), unless not feasible as determined by the investigator and discussed with the sponsor

Safety Run-in Cohort 1 and Phase 2 Cohort 1 (Ineligible (1L) Unfit acute myeloid leukemia (AML) Magrolimab + Venetoclax + Azacitidine):

* Newly diagnosed, previously untreated individuals with histological confirmation of AML by world health organization (WHO) criteria who are ineligible for treatment with a standard cytarabine and anthracycline induction regimen due to age, comorbidity, or other factors. Individuals must be considered ineligible for induction therapy defined by the following:

  * ≥ 75 years of age
  * ≥ 18 to 74 years of age with at least 1 of the following comorbidities:

    * Diffusing capacity of the lung of carbon monoxide ≤ 65% or forced expiratory volume in 1 second ≤ 65%
    * Left ventricular ejection fraction (LVEF) ≤ 50%
    * Creatinine clearance (CrCl) < 45 mL/min calculated by the Cockcroft-Gault formula or measured by 24 hours' urine collection
    * Any other comorbidity that the investigator judges to be incompatible with intensive chemotherapy that must be approved by the sponsor medical monitor before study enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or 3
* Individuals who have not received prior anti-leukemia therapy for AML (excluding hydroxyurea or oral etoposide), hypomethylating agent (HMA), low-dose cytarabine, and/or venetoclax. Individuals with prior myelodysplastic syndrome (MDS) cannot have received a prior HMA, venetoclax, or a chemotherapeutic agent. Other prior MDS therapies, including but not limited to lenalidomide, erythroid-stimulating agents, or similar red blood cell (RBC) -direct therapies, are allowed
* Individuals who have not received strong and/or moderate cytochrome P450 enzyme (CYP) 3A inducers (such as St. John's Wort) within 7 days prior to the initiation of study treatment
* Individuals who have not consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or starfruit within 3 days prior to the initiation of study treatment or are willing to discontinue consumption of these while receiving study drug
* Individuals without malabsorption syndrome or other conditions that preclude enteral route of administration

Safety Run-in Cohort 2 and Phase 2 Cohort 2 (Relapsed/refractory (R/R) AML Magrolimab+Mitoxantrone + Etoposide + Cytarabine (MEC)):

* Individuals with confirmation of AML by WHO criteria who are refractory to or have experienced first relapse after initial intensive chemotherapy. Note: Individuals who are relapsed after or are refractory to more than 1 line of anti-AML treatment are not eligible. Individuals who relapsed after undergoing stem cell transplant may be eligible.
* At least 2 weeks must have elapsed since any prior anti-leukemia agents. Note: Localized non-central nervous system (CNS) radiotherapy, hydroxyurea, and erythroid and/or myeloid growth factors are not criteria for exclusion
* ECOG performance status of 0 to 2
* Individuals with LVEF > 50%, lack of symptomatic congestive heart failure, or clinically significant cardiac arrhythmias
* Must not have been treated with trastuzumab within 7 months prior to the initiation of study treatment
* Individuals who have not previously received maximum cumulative doses of anthracyclines and anthracenediones
* Individuals without degenerative or toxic encephalopathies.
* Individuals who did not undergo hematopoietic SCT in the past 100 days, are not on immunosuppressive therapy post SCT in the 2 weeks prior to the first dose of study treatment, or have no active clinically significant graft-versus-host disease.

Safety Run-in Cohort 3 and Phase 2 Cohort 3 (Post-chemo Maintenance Magrolimab+CC-486):

* Individuals with histological confirmation of AML by WHO criteria who achieved a complete remission (CR) or CR with incomplete hematologic recovery (CRi) with presence of MRD (MRD positive by flow cytometry assay, defined as ≥ 0.1% detectable MRD) after intensive induction chemotherapy with or without consolidation therapy, prior to starting maintenance therapy for newly diagnosed AML, and who are not candidates for hematopoietic stem cell transplantation (SCT) within 1 year of achievement of initial remission
* ECOG performance status of 0 to 2
* Individuals without malabsorption syndrome or other conditions that preclude enteral route of administration

Key Exclusion Criteria:

* Positive serum pregnancy test
* Breastfeeding female
* Known hypersensitivity to any of the study drugs, the metabolites, or formulation excipient
* Individuals receiving any live virus vaccine within 4 weeks prior to initiation of study treatments
* Prior treatment with cluster of differentiation 47 (CD47) or signal regulatory protein alpha (SIRPα) -targeting agents
* Current participation in another interventional clinical trial
* Known inherited or acquired bleeding disorders
* Clinical suspicion of or documented active CNS involvement with AML
* Individuals who have acute promyelocytic leukemia
* Significant disease or medical conditions, as assessed by the investigator and sponsor, that would substantially increase the risk: benefit ratio of participating in the study. This includes, but is not limited to, acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, and congestive heart failure New York Heart Association Class III-IV
* Second malignancy, except MDS, treated basal cell or localized squamous skin carcinomas, localized prostate cancer, or other malignancies for which individuals are not on active anti-cancer therapies and have had no evidence of active malignancy for over 1 year. Previous hormonal therapy with luteinizing hormone-releasing hormone (LHRH) agonists for prostate cancer and treatment with bisphosphonates and receptor activator of nuclear factor kappa-B ligand (RANKL) inhibitors are not criteria for exclusion

  * Note: Individuals on maintenance therapy alone who have no evidence of active malignancy for at least ≥ 1 year are eligible.
* Known active or chronic hepatitis B or C infection or human immunodeficiency virus

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (21):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OU Health, Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Oxford University Hospitals NHS Foundation Trust, Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mannis GN, Abboud C, Daver NG, Guru Murthy GS, Wang ES, Bradley TJ, et al. Tolerability and Efficacy of Magrolimab Plus Mitoxantrone, Etoposide, and Cytarabine (MEC) in Patients with Acute Myeloid Leukemia (AML) Refractory/Relapsed (R/R) After Induction Chemotherapy (IC). European Hematology Association (EHA) 13-16 June 2024.
- [Derived] Mannis GN, Abboud CN, Daver NG, Murthy GSG, Wang ES, Bradley TJ, Yaghmour G, Vachhani P, Balasubramanian SK, Chua CC, Fong CY, Asch AS, Dong M, Li S, Bagheri T, Doshi P, Vyas P, Malki MMA. Phase 2 Multi-Arm Study of Magrolimab Combinations in Patients With Acute Myeloid Leukaemia. EJHaem. 2025 May 13;6(3):e70051. doi: 10.1002/jha2.70051. eCollection 2025 Jun. PMID 40364806
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-546-5920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 77 participants were screened.
Pre-assignment Details: Participants were enrolled at study sites in the United States, the United Kingdom and Australia.
  No participants were enrolled in Cohort 3, so, results are reported only for Cohorts 1 and 2.
  Due to limited number of participants enrolled, and because all participants were dosed with same dose of magrolimab, per prespecified analysis, data for Safety Run-in and Phase 2 Cohorts were combined in outcome measures (OMs) except DLT OM, for which data was collected only in Safety Run-in Cohorts
Groups:
- Safety Run-in Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine: Participants in Safety Run-in Cohort 1 with untreated AML who were unfit for chemotherapy received the recommended dose of magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then every week (QW) x 5 doses; 30 mg/kg over 2 hours every 2 weeks (Q2W) beginning 1 week after the 5 weekly 30 mg/kg dose, intravenously (IV) in 28-day cycles.
  Participants also received azacitidine 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9, subcutaneously (SC) or IV, along with venetoclax oral tablets, 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Days 3 to 28 of Cycle 1, 400 mg on Days 1 to 28 in Cycle 2 and consecutive cycles for every 28-day cycle. The treatment duration was up to a maximum of 1.7 years.
- Safety Run-in Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine): Participants in Safety Run-in Cohort 2 with R/R AML received the recommended dose of magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 doses; 30 mg/kg Q2W beginning 1 week after the 5 weekly 30 mg/kg dose, IV up to 1.7 years. Participants also received MEC: mitoxantrone 8 mg/m^2 IV, etoposide 100 mg/m^2 IV and cytarabine 1000 mg/m^2 IV on Days 1 to 5 for three 28-day cycles.
- Safety Run-in Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486; Phase 2 Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486: Participants with AML who achieved CR or CRi with intensive induction chemotherapy were to receive magrolimab along with CC-486. However, the cohort was closed before any participants could join, so no doses were given.
- Phase 2 Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine: Participants in Phase 2 Cohort 1 with untreated AML who were unfit for chemotherapy received the recommended dose of magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then every week (QW) x 5 doses; 30 mg/kg over 2 hours every 2 weeks (Q2W) beginning 1 week after the 5 weekly 30 mg/kg dose, intravenously (IV) in 28-day cycles.
  Participants also received azacitidine 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9, subcutaneously (SC) or IV, along with venetoclax oral tablets, 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Days 3 to 28 of Cycle 1, 400 mg on Days 1 to 28 in Cycle 2 and consecutive cycles for every 28-day cycle. The treatment duration was up to a maximum of 1.7 years.
- Phase 2 Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine): Participants in Phase 2 Cohort 2 with R/R AML received the recommended dose of magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 doses; 30 mg/kg Q2W beginning 1 week after the 5 weekly 30 mg/kg dose, IV up to 1.7 years. Participants also received MEC: mitoxantrone 8 mg/m^2 IV, etoposide 100 mg/m^2 IV and cytarabine 1000 mg/m^2 IV on Days 1 to 5 for three 28-day cycles.
Period: Safety Run-in Period
Arm/Group | Safety Run-in Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Safety Run-in Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Safety Run-in Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486 | Phase 2 Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Phase 2 Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Phase 2 Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Started | 7 | 6 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 6 | 0 | 0 | 0 | 0
Not completed — Death | 5 | 6 | 0 | 0 | 0 | 0
Period: Phase 2 Period
Arm/Group | Safety Run-in Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Safety Run-in Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Safety Run-in Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486 | Phase 2 Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Phase 2 Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Phase 2 Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Started | 0 | 0 | 0 | 11 | 30 | 0
Completed | 0 | 0 | 0 | 4 | 9 | 0
Not Completed | 0 | 0 | 0 | 7 | 21 | 0
Not completed — Death | 0 | 0 | 0 | 5 | 18 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The All-Enrolled Analysis Set included all participants who received a study patient identification (ID) number in the study after screening.
  Per pre-specified analysis, the arms for both Cohorts 1 and 2 for Safety Run-in and Phase 2 periods were combined for analysis.
Groups:
- Safety Run-in Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine: Participants in Safety Run-in Cohort 1 with untreated AML who were unfit for chemotherapy received magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then every week (QW) x 5 doses; 30 mg/kg over 2 hours every 2 weeks (Q2W) beginning 1 week after the 5 weekly 30 mg/kg dose, intravenously (IV) for 28 days.
  Participants also received azacitidine 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9, subcutaneously (SC) or IV, along with venetoclax oral tablets, 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Days 3 to 28 of Cycle 1, 400 mg on Days 1 to 28.
- Safety Run-in Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine): Participants in Safety Run-in Cohort 2 with R/R AML received magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 doses; 30 mg/kg Q2W beginning 1 week after the 5 weekly 30 mg/kg dose, IV for 28 days. Participants also received MEC: mitoxantrone 8 mg/m^2 IV, etoposide 100 mg/m^2 IV and cytarabine 1000 mg/m^2 IV on Days 1 to 5 for 28 days.
- Phase 2 Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine: Participants in Phase 2 Cohort 1 with untreated AML who were unfit for chemotherapy received the recommended dose of magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 doses; 30 mg/kg over 2 hours Q2W beginning 1 week after the 5 weekly 30 mg/kg dose, IV in 28-day cycles.
  Participants also received azacitidine 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9, SC or IV, along with venetoclax oral tablets, 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Days 3 to 28 of Cycle 1, 400 mg on Days 1 to 28 in Cycle 2 and consecutive cycles for every 28-day cycle. The treatment duration was up to a maximum of 1.7 years.
- Total: Total of all reporting groups
Arm/Group | Safety Run-in Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Safety Run-in Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Phase 2 Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Phase 2 Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Total
Number analyzed (Participants) | 7 | 6 | 11 | 30 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (8.6) | 47 (14.9) | 72 (4.3) | 51 (14.0) | 58 (16.1)
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: < 50 Years | 0 | 3 | 0 | 13 | 16
  Age, Categorical: >= 50 - < 75 Years | 3 | 3 | 9 | 17 | 32
  Age, Categorical: >= 75 Years | 4 | 0 | 2 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 5 | 14 | 23
  Male | 4 | 5 | 6 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 6 | 10
  Not Hispanic or Latino | 6 | 3 | 11 | 23 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2 | 4
  White | 7 | 2 | 9 | 23 | 41
  More than one race | 0 | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate (Cohorts 1 and 2)
Description: CR rate was the percentage of participants who achieved CR (CR without minimal residual disease (CRMRD-) or complete remission with positive or unknown minimal residual disease (CRMRD+/unk)) as determined by the investigator based on prespecified criteria while on study prior to initiation of any new anti-cancer therapy. CRMRD- and CRMRD+/unk were defined as neutrophils >1.0 ×10^9/L; platelets >100 × 10^9/L and <5% bone marrow blasts. Absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease. CRMRD- status as determined using multiparameter flow cytometry with a sensitivity of < 0.1%. Assessment of leukemia response in participants with acute myeloid leukemia (AML) were conducted based on the European Leukemia Net (ELN) recommendations for AML.
  Percentages were rounded-off. Clopper-Pearson method was used for outcome measure analysis.
Time Frame: Up to 2 years
Population: The Full Analysis Set included all enrolled participants who received at least 1 dose of any study treatment, with treatment group designated according to the assigned treatment.
  Per pre-specified analysis, the arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis as participants in Cohorts 1 and 2 received the same dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine: Participants in Safety Run-in and Phase 2 Cohorts in Cohort 1 with untreated AML who were unfit for chemotherapy received the recommended dose of magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then every week (QW) x 5 doses; 30 mg/kg over 2 hours every 2 weeks (Q2W) beginning 1 week after the 5 weekly 30 mg/kg dose, intravenously (IV) in 28-day cycles.
  Participants also received azacitidine 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9, subcutaneously (SC) or IV, along with venetoclax oral tablets, 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Days 3 to 28 of Cycle 1, 400 mg on Days 1 to 28 in Cycle 2 and consecutive cycles for every 28-day cycle. The treatment duration was up to a maximum of 1.7 years.
- Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine): Participants in Safety Run-in and Phase 2 Cohorts in Cohort 2 with R/R AML received the recommended dose of magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 doses; 30 mg/kg Q2W beginning 1 week after the 5 weekly 30 mg/kg dose, IV up to 1.7 years. Participants also received MEC: mitoxantrone 8 mg/m^2 IV, etoposide 100 mg/m^2 IV and cytarabine 1000 mg/m^2 IV on Days 1 to 5 for three 28-day cycles.
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine)
Number analyzed (Participants) | 18 | 36
percentage of participants | 38.9 [17.3 to 64.3] | 25 [12.1 to 42.2]
Statistical Analysis 1: Comparison: Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine); Test type: Superiority; p = 0.1794, One Group Chi-Square test; The p-value was based on one group Chi-Square test for the null hypothesis CR rate was 0.19 at one-sided alpha of 0.1 in Cohort 2

2. Primary Outcome: Minimal Residual Disease Negative Complete Remission Rate (Cohort 3)
Description: The minimal residual disease (MRD) negative CR rate was defined as the percentage of participants who maintain CR as determined by the investigator based on prespecified criteria and reach MRD negative disease status on 2 consecutive bone marrow assessments, as determined using multiparameter flow cytometry with a sensitivity of < 0.1% while on study prior to initiation of any new anti-AML therapy. Assessment of leukemia response in participants with AML were conducted based on the ELN recommendations for AML. CR was defined in outcome measure #1.
Time Frame: Up to 2 years
Population: As no participants were enrolled in Cohort 3, data for Cohort 3 were not collected for this outcome measure.
Groups:
- Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486: Participants with AML who achieved CR or CRi with intensive induction chemotherapy were to receive magrolimab along with CC-486. However, the cohort was closed before any participants could join, so no doses were given.
Arm/Group | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 0

3. Primary Outcome: Percentage of Participants Experiencing Dose-limiting Toxicities (DLTs) (Safety Run-in Cohorts 1, 2 and 3)
Description: DLTs were defined as any Grade 4 or higher hematologic toxicity or Grade 3 or higher nonhematologic toxicity (that had worsened in severity from pretreatment baseline) during the 4-week DLT assessment period and was related to magrolimab or magrolimab combination.
Time Frame: Up to 28 days
Population: The DLT Evaluable Analysis Set included all participants in the Safety Analysis Set who were enrolled in the Safety Run-in cohorts, have safety assessments through the protocol-specified DLT assessment window (first 4 weeks of study dosing, inclusive), and fulfill the criteria for evaluation for DLT specified in the protocol.
  As no participants were enrolled in Cohort 3, data for Cohort 3 were not collected for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 6 | 6 | 0
percentage of participants | 0 | 0 |

4. Primary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) (Cohorts 1, 2 and 3)
Description: TEAEs were defined as any AEs with an onset date on or after the study drug start date and no later than 70 days after the study drug last dosing date or the day before initiation of new anticancer therapy including SCT, whichever comes first. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
  Percentages were rounded-off.
Time Frame: First dose date up to 1.7 years plus 70 days
Population: The Safety Analysis Set included all participants who received at least 1 dose of study treatment, with treatment assignments designated according to the actual treatment received.
  Per pre-specified analysis, the arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis as participants in Cohorts 1 and 2 received the same dose.
  As no participants were enrolled in Cohort 3, data for Cohort 3 were not collected for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 18 | 36 | 0
percentage of participants | 100 | 97.2 |

5. Primary Outcome: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities (Cohorts 1, 2 and 3)
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 70 days or the day before initiation of any new anticancer therapy including SCT, whichever comes first. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment emergent.
  Percentages were rounded-off.
Time Frame: First dose date up to 1.7 years plus 70 days
Population: Participants in the Safety Analysis Set were analyzed. Per pre-specified analysis, the arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis as participants in Cohorts 1 and 2 received the same dose.
  As no participants were enrolled in Cohort 3, data for Cohort 3 were not collected for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 18 | 36 | 0
percentage of participants | 100 | 97.2 |

6. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was the percentage of participants who achieved CR (CRMRD- or CRMRD+/unk), CRi, CRh, PR, or MLFS as per investigator based on prespecified criteria before starting any new anti-AML therapy (including SCT). CRi and CRh were defined as neutrophils >0.5 x 10^9/L, platelets > 50 x 10^9/L (except residual neutropenia (<1.0 × 10^9/L) or thrombocytopenia (<100 × 109/L) for CRi) and bone marrow blasts <5%; Absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease. PR: Neutrophils >1.0 x 10^9/L, platelets >100 x 10^9/L, bone marrow blasts reduced to 5%-25%, and a ≥50% reduction from baseline. Blasts <5% with Auer rods may also be considered a PR. MLFS: Bone marrow blasts <5%, absence of circulating blasts or Auer rods, no extramedullary disease, marrow should not merely be "aplastic"; at least 200 cells or 10% cellularity, and no requirement for hematologic recovery. CR was defined in outcome measure #1.
  Percentages were rounded-off.
Time Frame: Up to 2 years
Population: Participants in the Full Analysis Set were analyzed. Clopper-Pearson exact method was used in outcome measure analysis.
  Per pre-specified analysis, the arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis as participants in Cohorts 1 and 2 received the same dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine)
Number analyzed (Participants) | 18 | 36
percentage of participants | 66.7 [41.0 to 86.7] | 38.9 [23.1 to 56.5]

7. Secondary Outcome: Complete Remission or Complete Remission With Partial Hematologic Recovery Rate (CR/CRh) (Cohorts 1 and 2)
Description: CR/CRh rate was the percentage of participants who achieved CR (CRMRD- or CRMRD+/unk) or CRh as determined by the investigator based on prespecified criteria while on study prior to initiation of any new anti-AML therapy (including SCT). CR was defined in outcome measure 1. CRh was defined in outcome measure 6. Percentages were rounded-off. Clopper-Pearson exact method was used in outcome measure analysis.
Time Frame: Up to 2 years
Population: Participants in the Full Analysis Set were analyzed. Per pre-specified analysis, the arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis as participants in Cohorts 1 and 2 received the same dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine)
Number analyzed (Participants) | 18 | 36
percentage of participants | 44.4 [21.5 to 69.2] | 30.6 [16.3 to 48.1]

8. Secondary Outcome: Duration of Response (DOR) (Cohorts 1 and 2)
Description: DOR was measured from the time assessment criteria that were met for CR (CRMRD- or CRMRD+/unk), CRi, CRh, PR, or MLFS, whichever was first recorded, until the first date of AML relapse, progressive disease, or death (including assessments post SCT). Participants who were not observed to have a relapse, progressive disease, or death were censored at the date of their last response assessment. For participants who started taking new anti-AML therapies (except SCT and post SCT maintenance treatment) before relapse/PD/death, duration of response were censored at the last response assessment before the initiation of the new anti-AML therapies.CR was defined in outcome measure #1. CRi, CRh, PR, or MLFS were defined in outcome measure #6.
  Kaplan-Meier (KM) estimates were used in outcome measure analysis.
Time Frame: Up to 2 years
Population: Participants in the Full Analysis Set who achieved overall response were analyzed. Per pre-specified analysis, the arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis as participants in Cohorts 1 and 2 received the same dose.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine)
Number analyzed (Participants) | 12 | 14
months | 15.9 [2.2 to NA] — Upper limit of confidence interval (CI) was not estimable due to insufficient number of participants with events. | 8.7 [6.3 to NA] — Upper limit of confidence interval (CI) was not estimable due to insufficient number of participants with events.

9. Secondary Outcome: Duration of Complete Remission (DCR) (Cohorts 1 and 2)
Description: DCR was measured from the time the assessment criteria were first met for CR (CRMRD- or CRMRD+/unk) until the first date of AML relapse or death (including assessments post SCT). Participants who were not observed to have a relapse, progressive disease, or death were censored at the date of their last response assessment. For participants who started taking new anti-AML therapies (except SCT and post SCT maintenance treatment) before relapse/PD/death, duration of response were censored at the last response assessment before the initiation of the new anti-AML therapies. CR was defined in outcome measure #1.
  KM estimates were used in outcome measure analysis.
Time Frame: Up to 2 years
Population: Participants in the Full Analysis Set who achieved CR were analyzed. Per pre-specified analysis, the arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis as participants in Cohorts 1 and 2 received the same dose.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine)
Number analyzed (Participants) | 7 | 9
months | 15.9 [6.7 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events. | 8.7 [2.3 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events.

10. Secondary Outcome: Duration of CR/CRi (Cohorts 1 and 2)
Description: Duration of CR/CRi was measured from the time the assessment criteria were first met for CR (CRMRD- or CRMRD+/unk) or CRi until the first date of AML relapse or death (including assessments post SCT). Participants who were not observed to have a relapse, progressive disease, or death were censored at the date of their last response assessment. For participants who started taking new anti-AML therapies (except SCT and post SCT maintenance treatment) before relapse/PD/death, duration of response were censored at the last response assessment before the initiation of the new anti-AML therapies. CR was defined in outcome measure #1. CRi was defined in outcome measure #6.
  KM estimates were used in outcome measure analysis.
Time Frame: Up to 2 years
Population: Participants in the Full Analysis Set who achieved CR/CRi were analyzed. Per pre-specified analysis, the arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis as participants in Cohorts 1 and 2 received the same dose.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine)
Number analyzed (Participants) | 9 | 11
months | 15.9 [3.9 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events. | 8.7 [2.3 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events.

11. Secondary Outcome: Duration of CR/CRh (Cohorts 1 and 2)
Description: Duration of CR/CRh was measured from the time the assessment criteria are first met for CR (CRMRD- or CRMRD+/unk) or CRh until the first date of AML relapse or death (including assessments post SCT). Participants who were not observed to have a relapse, progressive disease, or death were censored at the date of their last response assessment. For participants who started taking new anti-AML therapies (except SCT and post SCT maintenance treatment) before relapse/PD/death, duration of response were censored at the last response assessment before the initiation of the new anti-AML therapies. CR was defined in outcome measure #1. CRh was defined in outcome measure #6.
  KM estimates were used in outcome measure analysis.
Time Frame: Up to 2 years
Population: Participants in the Full Analysis Set who achieved CR/CRh were analyzed. Per pre-specified analysis, the arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis as participants in Cohorts 1 and 2 received the same dose.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine)
Number analyzed (Participants) | 8 | 11
months | 15.9 [6.7 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events. | 8.7 [2.3 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events.

12. Secondary Outcome: Event-Free Survival (EFS) (Cohorts 1 and 2)
Description: EFS was defined as the time from the date of the first dose of study treatment to the earliest date of documented relapse from CR, treatment failure (defined as failure to achieve CR during the response assessment window (the first treatment dosing date until before the fifth cycle of magrolimab + venetoclax + azacitidine in Cohort 1 and the first treatment dosing date until before the third cycle of magrolimab + MEC in Cohort 2), or death from any cause within the response assessment window. Response assessments post SCT were included in the analysis. Deaths post SCT or new anti-AML therapies (except SCT and post SCT maintenance) were included. Those who were not observed to have one of these events during the study were censored at the date of their last response assessment during the study. Day 1 of treatment was assigned as the event date for participants with treatment failure. CR was defined in outcome measure #1.
  KM estimates were used in outcome measure analysis.
Time Frame: Up to 2 years
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine)
Number analyzed (Participants) | 18 | 36
months | 3.8 [0.0 to 16.8] | 0.0 [NA to NA] — Upper and lower limits of the CI could not be estimated due to a limitation in the Kaplan-Meier model, as EFS values were below the level of quantification for this outcome measure.

13. Secondary Outcome: Relapse-Free Survival (RFS) Rate (Cohort 3)
Description: RFS was defined as the time from the first dose of study treatment until the first date of AML relapse or death from any cause, whichever came first.
Time Frame: Up to 2 years
Population: As no participants were enrolled in Cohort 3, data for Cohort 3 were not collected for this outcome measure.
Arm/Group | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 0

14. Secondary Outcome: MRD Negative CR/CRi Rate (Cohort 3)
Description: MRD negative CR/CRi rate was defined as the percentage of participants who maintained CR/CRi as determined by the investigator based on prespecified criteria and reach MRD negative disease status on 2 consecutive bone marrow assessments as determined using multiparameter flow cytometry with a sensitivity of < 0.1% while on study prior to initiation of any new anti-AML therapy. CR was defined in outcome measure #1. CRi was defined in outcome measure #6.
Time Frame: Up to 2 years
Population: As no participants were enrolled in Cohort 3, data were not collected for this outcome measure.
Arm/Group | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 0

15. Secondary Outcome: Duration of Minimal Residual Disease Negative Complete Remission (Cohort 3)
Description: Duration of MRD negative CR was measured from the time the participant achieved MRD-negative status and maintained CR until the first date of AML relapse, loss of MRD negative status, or death (including assessments post SCT). CR was defined in outcome measure #1.
Time Frame: Up to 2 years
Population: As no participants were enrolled in Cohort 3, data for Cohort 3 were not collected for this outcome measure.
Arm/Group | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 0

16. Secondary Outcome: Duration of MRD Negative CR/CRi (Cohort 3)
Description: Duration of MRD negative CR/CRi was measured from the time the participant achieved MRD-negative status (first of the 2 consecutive MRD negative bone marrow assessments) and maintained CR/CRi until the first date of AML relapse, loss of MRD negative status, or death (including assessments post SCT). CR was defined in outcome measure #1. CRi was defined in outcome measure #6.
Time Frame: Up to 2 years
Population: As no participants were enrolled in Cohort 3, data were not collected for this outcome measure.
Arm/Group | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 0

17. Secondary Outcome: Overall Survival (OS) (Cohorts 1, 2 and 3)
Description: OS was measured from the date of the first dose of study treatment to the date of death from any cause. Those who were not observed to die during the study were censored at last date they were known to be alive.
  KM estimates were used in outcome measure analysis.
Time Frame: Up to 2 years
Population: Participants in the Full Analysis Set were analyzed. Per pre-specified analysis, the arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis as participants in Cohorts 1 and 2 received the same dose.
  As no participants were enrolled in Cohort 3, data for Cohort 3 were not collected for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 18 | 36 | 0
months | 15.3 [3.1 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events. | 10.5 [7.1 to 15.4] |

18. Secondary Outcome: Red Blood Cell (RBC) Transfusion Independence Rate (Cohorts 1, 2 and 3)
Description: RBC transfusion independence rate was the percentage of participants who had a 56-day or longer period with no RBC or whole blood transfusion at any time between the date of the first dose and discontinuation of study treatment among all participants who were RBC transfusion-dependent at baseline. RBC transfusion independence rate was reported as 2 categories:
  1. Conversion rate: Participants who received an RBC or whole blood transfusion within the 28 days prior to the first dose of study treatment, and were RBC transfusion-independent post-baseline.
  2. Maintenance rate: Participants who were RBC transfusion independent at baseline and maintained it post-baseline.
  Percentages were rounded-off. Clopper-Pearson method were used in outcome measure analysis.
Time Frame: Up to 2 years
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 18 | 36 | 0
percentage of participants
  RBC Transfusion Independence (Conversion) Rate: number analyzed (Participants) | 13 | 26 | 0
  RBC Transfusion Independence (Conversion) Rate | 30.8 [9.1 to 61.4] | 3.8 [0.1 to 19.6] |
  RBC Transfusion Independence (Maintenance) Rate: number analyzed (Participants) | 5 | 10 | 0
  RBC Transfusion Independence (Maintenance) Rate | 60.0 [14.7 to 94.7] | 20.0 [2.5 to 55.6] |

19. Secondary Outcome: Platelet Transfusion Independence Rate (Cohorts 1, 2 and 3)
Description: Platelet transfusion independence rate was the percentage of participants who had a 56-day or longer period with no platelet transfusions at any time between the date of the first dose and discontinuation of study treatment among all participants who were platelet transfusion-dependent at baseline. Platelet transfusion independence rate was reported as 2 categories:
  1. Conversion rate: Participants who received an platelet transfusion within 28 days prior to the first dose of study treatment,
  2. Maintenance rate: Participants who were platelet transfusion independent at baseline and maintained it post-baseline.
  Percentages were rounded-off. Clopper-Pearson method were used in outcome measure analysis.
Time Frame: Up to 2 years
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 18 | 36 | 0
percentage of participants
  Platelet Transfusion Independence (Conversion) Rate: number analyzed (Participants) | 3 | 23 | 0
  Platelet Transfusion Independence (Conversion) Rate | 0.0 [0.0 to 70.8] | 8.7 [1.1 to 28.0] |
  Platelet Transfusion Independence (Maintenance) Rate: number analyzed (Participants) | 15 | 13 | 0
  Platelet Transfusion Independence (Maintenance) Rate | 60.0 [32.3 to 83.7] | 7.7 [0.2 to 36.0] |

20. Secondary Outcome: Plasma Concentration of Magrolimab in Combination With Anti-leukemia Therapy (Cohorts 1, 2 and 3)
Time Frame: Cohort 1: Predose: Days 1, 8, 29, 57, 113, 169, 253 and 337; Cohort 2: Days 1, 8, 29 and 57
Population: The Pharmacokinetic Analysis Set included all enrolled participants who received at least 1 dose of magrolimab and 1 measurable (non-below the limit of quantitation numeric values) post-treatment serum concentration of magrolimab. Participants with available data were analyzed. Per pre-specified analysis, arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis.
  As no participants were enrolled in Cohort 3, data for Cohort 3 were not collected for this outcome measure.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 13 | 25 | 0
μg/mL
  Predose: Day 1 | 0.0 (0.0) | 0.0 (0.0) |
  Predose: Day 8: number analyzed (Participants) | 11 | 25 | 0
  Predose: Day 8 | 0.0 (0.0) | 0.0 (0.0) |
  Predose: Day 29: number analyzed (Participants) | 10 | 20 | 0
  Predose: Day 29 | 376 (271) | 507 (272) |
  Predose: Day 57: number analyzed (Participants) | 8 | 9 | 0
  Predose: Day 57 | 1050 (925) | 824 (581) |
  Predose: Day 113: number analyzed (Participants) | 3 | 0 | 0
  Predose: Day 113 | 648 (314) |  |
  Predose: Day 169: number analyzed (Participants) | 2 | 0 | 0
  Predose: Day 169 | 592 (371) |  |
  Predose: Day 253: number analyzed (Participants) | 2 | 0 | 0
  Predose: Day 253 | 178 (166) |  |
  Predose: Day 337: number analyzed (Participants) | 1 | 0 | 0
  Predose: Day 337 | 337 (NA) — Standard deviation could not be calculated for 1 participant. |  |

21. Secondary Outcome: Percentage of Participants With Anti-Magrolimab Antibodies (Cohorts 1 and 2)
Description: Percentages were rounded-off.
Time Frame: Up to 2 years
Population: The Immunogenicity Analysis Set included all enrolled participants who received at least 1 dose of magrolimab and have at least 1 reported anti-magrolimab antibody test result. Participants with post-baseline data were analyzed.
  Per pre-specified analysis, arms for Cohorts 1 and 2 for Safety Run-in and Phase 2 were combined for analysis as participants in Cohorts 1 and 2 received same dose.
  As no participants were enrolled in Cohort 3, data for Cohort 3 were not collected.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 14 | 26 | 0
percentage of participants | 0 | 0 |

22. Secondary Outcome: Levels of Anti-Magrolimab Antibodies (Cohorts 1 and 2)
Time Frame: Up to 2 years
Population: Participants in the Immunogenicity Analysis Set with post-baseline data were analyzed. Per Specified analysis, the arms for both Cohorts 1 and 2 for Safety Run-in and Phase 2 periods were combined for analysis.
  As no participants were enrolled in Cohort 3, data for Cohort 3 were not collected for this outcome measure.
Measure: Number; unit: titer
Arm/Group | Cohort 1 (1L, Unfit AML): Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Cohort 3 (Post-Chemo Maintenance): Magrolimab + CC-486
Number analyzed (Participants) | 14 | 26 | 0
titer | NA — ADA levels could not be analyzed as there were no positive samples available for analysis. | NA — ADA levels could not be analyzed as there were no positive samples available for analysis. |

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 2 years; Adverse events: Up to 1.7 years plus 70 days
Description: All-cause mortality: The All-Enrolled Analysis Set included all participants who received a study patient identification (ID) number in the study after screening.
  Adverse events: The Safety Analysis Set included all participants who received at least 1 dose of study treatment, with treatment assignments designated according to the actual treatment received.
  As no participants were enrolled in Cohort 3, data for adverse events were reported only for Cohorts 1 and 2.
Groups:
- Cohort 1 (1L, Unfit AML): Safety Run-In Cohort: Magrolimab + Venetoclax + Azacitidine: Participants in Safety Run-in Cohort in Cohort 1 with untreated AML who were unfit for chemotherapy received magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then every week (QW) x 5 doses; 30 mg/kg over 2 hours every 2 weeks (Q2W) beginning 1 week after the 5 weekly 30 mg/kg dose, intravenously (IV) for 28 days.
  Participants also received azacitidine 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9, subcutaneously (SC) or IV, along with venetoclax oral tablets, 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Days 3 to 28 of Cycle 1, 400 mg on Days 1 to 28.
- Cohort 2 (R/R AML): Safety Run-In Cohort: Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine): Participants in Safety Run-in Cohort in Cohort 2 with R/R AML received magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 doses; 30 mg/kg Q2W beginning 1 week after the 5 weekly 30 mg/kg dose, IV for 28 days. Participants also received MEC: mitoxantrone 8 mg/m^2 IV, etoposide 100 mg/m^2 IV and cytarabine 1000 mg/m^2 IV on Days 1 to 5 for 28 days.
- Cohort 1 (1L, Unfit AML): Phase 2 Cohort: Magrolimab + Venetoclax + Azacitidine: Participants in Phase 2 Cohort in Cohort 1 with untreated AML who were unfit for chemotherapy received the recommended dose of magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 doses; 30 mg/kg over 2 hours Q2W beginning 1 week after the 5 weekly 30 mg/kg dose, IV in 28-day cycles.
  Participants also received azacitidine 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9, SC or IV, along with venetoclax oral tablets, 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Days 3 to 28 of Cycle 1, 400 mg on Days 1 to 28 in Cycle 2 and consecutive cycles for every 28-day cycle. The treatment duration was up to a maximum of 1.7 years.
- Cohort 2 (R/R AML): Phase 2: Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine): Participants in Phase 2 Cohort in Cohort 2 with R/R AML received the recommended dose of magrolimab, 1 mg/kg on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 doses; 30 mg/kg Q2W beginning 1 week after the 5 weekly 30 mg/kg dose, IV up to 1.7 years. Participants also received MEC: mitoxantrone 8 mg/m^2 IV, etoposide 100 mg/m^2 IV and cytarabine 1000 mg/m^2 IV on Days 1 to 5 for three 28-day cycles.
Arm/Group | Cohort 1 (1L, Unfit AML): Safety Run-In Cohort: Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Safety Run-In Cohort: Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) | Cohort 1 (1L, Unfit AML): Phase 2 Cohort: Magrolimab + Venetoclax + Azacitidine | Cohort 2 (R/R AML): Phase 2: Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine)
All-Cause Mortality (participants affected / at risk) | 5/7 | 6/6 | 5/11 | 19/30
Serious Adverse Events (participants affected / at risk) | 7/7 | 3/6 | 11/11 | 18/30
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 11/11 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (1L, Unfit AML): Safety Run-In Cohort: Magrolimab + Venetoclax + Azacitidine (N=7) | Cohort 2 (R/R AML): Safety Run-In Cohort: Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) (N=6) | Cohort 1 (1L, Unfit AML): Phase 2 Cohort: Magrolimab + Venetoclax + Azacitidine (N=11) | Cohort 2 (R/R AML): Phase 2: Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 6
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 1
Infusion related hypersensitivity reaction (Immune system disorders) | 0 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 1 | 6
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Testicular abscess (Infections and infestations) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Lacunar stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (1L, Unfit AML): Safety Run-In Cohort: Magrolimab + Venetoclax + Azacitidine (N=7) | Cohort 2 (R/R AML): Safety Run-In Cohort: Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) (N=6) | Cohort 1 (1L, Unfit AML): Phase 2 Cohort: Magrolimab + Venetoclax + Azacitidine (N=11) | Cohort 2 (R/R AML): Phase 2: Magrolimab + MEC (Mitoxantrone + Etoposide + Cytarabine) (N=30)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 6 | 14
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 12
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 2
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 3
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 2 | 4
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 3
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0
Vitreous degeneration (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 4 | 9
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 6 | 10
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2 | 4
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 0 | 5
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 7 | 14
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 4
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 7
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 10
Asthenia (General disorders) | 1 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 2 | 1
Chills (General disorders) | 1 | 2 | 2 | 6
Fatigue (General disorders) | 3 | 2 | 4 | 9
Injection site rash (General disorders) | 0 | 0 | 1 | 1
Localised oedema (General disorders) | 0 | 2 | 0 | 2
Malaise (General disorders) | 0 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 3
Oedema peripheral (General disorders) | 2 | 1 | 3 | 5
Pain (General disorders) | 0 | 1 | 2 | 2
Pyrexia (General disorders) | 1 | 3 | 6 | 16
Thirst (General disorders) | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic infarction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 3
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 1 | 1 | 0 | 3
Device related bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 2 | 3
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis fungal (Infections and infestations) | 0 | 2 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 2
Trichosporon infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 3
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 3 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 0 | 1 | 6
Blood bilirubin unconjugated increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1 | 0
Haptoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 3 | 5
Platelet count decreased (Investigations) | 3 | 3 | 6 | 7
Urine output decreased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 2 | 8
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 3 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4 | 4 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 1 | 3 | 11
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 3
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 3 | 4
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 3
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 3 | 13
Lethargy (Nervous system disorders) | 0 | 1 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 2 | 0
Thrombosis in device (Product Issues) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 3 | 3
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 2 | 2
Insomnia (Psychiatric disorders) | 2 | 2 | 4 | 7
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0
Sleep terror (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 2
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 2
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 3 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 2 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 3 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 5
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Embolism venous (Vascular disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 3 | 2
Hypotension (Vascular disorders) | 1 | 1 | 3 | 6
Jugular vein distension (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT04778410/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT04778410/SAP_001.pdf